CLINICAL TRIAL: NCT02945007
Title: A Phase 1, Open-label, Randomized Crossover Study, in Healthy Adult Subjects to Assess the Relative Oral Bioavailability of a Single 500-mg Dose of JNJ-53718678 Administered as (an) Oral Concept Formulation(s) Compared to the Current Oral Solution and to Assess the Effect of Food on the Pharmacokinetics of (an) Oral Concept Formulation(s)
Brief Title: A Study to Assess the Relative Oral Bioavailability of a Single Dose of JNJ-53718678 Administered as Oral Concept Formulation Compared to the Current Oral Solution and to Assess the Effect of Food on the Pharmacokinetics of Oral Concept Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108212; 2016-002665-59 (EudraCT Number); 53718678RSV1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-53718678

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- JNJ-53718678: PART 1 (Experimental): Participants will receive a single dose of JNJ-53718678 500 mg under fasted conditions on day 1 for treatment A (solution) and B (novel concept formulation 1), and under fed condition for treatment C (novel concept formulation 1).
  Interventions: Drug: JNJ-53718678
- JNJ-53718678: PART 2 (Experimental): Participants will receive a single dose of JNJ-53718678 500 mg under fasted conditions on day 1 for treatment A (solution) and D (novel concept formulation 2), and under fed condition for treatment E (novel concept formulation 2).
  Part 2 of the study is optional and might be performed depending on the availability of concept formulations and the result of previous part.
  Interventions: Drug: JNJ-53718678
- JNJ-53718678: PART 3 (Experimental): Participants will receive a single dose of JNJ-53718678 500 mg under fasted conditions on day 1 for treatment A (solution) and F (novel concept formulation 3), and under fed condition for treatment G (novel concept formulation 3).
  Part 3 of the study is optional and might be performed depending on the availability of concept formulations and the result of previous part.
  Interventions: Drug: JNJ-53718678
- JNJ-53718678: PART 4 (Experimental): Participants will receive a single dose of JNJ-53718678 500 mg under fasted conditions on day 1 for treatment A (solution) and H (novel concept formulation 4), and under fed condition for treatment I (novel concept formulation 4).
  Part 4 of the study is optional and might be performed depending on the availability of concept formulations and the result of previous part.
  Interventions: Drug: JNJ-53718678
- JNJ-53718678: PART 5 (Experimental): Participants will receive a single dose of JNJ-53718678 500 mg under fasted conditions on day 1 for treatment A (solution) and J (novel concept formulation 5), and under fed condition for treatment K (novel concept formulation 5).
  Part 5 of the study is optional and might be performed depending on the availability of concept formulations and the result of previous part.
  Interventions: Drug: JNJ-53718678
- JNJ-53718678: PART 6 (Experimental): Participants will receive a single dose of JNJ-53718678 500 mg under fasted conditions on day 1 for treatment A (solution) and L (novel concept formulation 6), and under fed condition for treatment M (novel concept formulation 6).
  Part 6 of the study is optional and might be performed depending on the availability of concept formulations and the result of previous part.
  Interventions: Drug: JNJ-53718678
- JNJ-53718678: PART 7 (Experimental): Participants will receive a single dose of JNJ-53718678 500 mg under fasted conditions on day 1 for treatment A (solution) and N (novel concept formulation 7), and under fed condition for treatment O (novel concept formulation 7).
  Part 7 of the study is optional and might be performed depending on the availability of concept formulations and the result of previous part.
  Interventions: Drug: JNJ-53718678
- JNJ-53718678: PART 8 (Experimental): Participants will receive a single dose of JNJ-53718678, 500 mg oral solution under fasted or fed conditions on day 1 for treatment A and P (oral concept formulation 1, 2, 3, 4, 5, 6 or 7) and under fed conditions for treatment Q (oral concept formulation 1, 2, 3, 4, 5, 6 or 7).
  Part 8 of the study is optional, might be performed, depending on the interim results of prior parts. One of the concept formulations might be re-evaluated under different feeding conditions.
  Interventions: Drug: JNJ-53718678

INTERVENTIONS:
Drug: JNJ-53718678 — Participants will receive JNJ-53718678 under fed or fasted conditions.

SUMMARY:
The purpose of this study is to assess the relative bioavailability of 1 to 3 concept formulations of JNJ-53718678 compared to the currently existing oral solution, and to assess the effect of food on the bioavailability of 1 to 3 oral concept formulations of JNJ-53718678 when administered as a single oral dose of 500 milligram (mg) in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* At Screening, a female participant must be of non-childbearing potential as defined in the protocol
* Female participants must have a negative serum beta human chorionic gonadotropin (beta-hCG) pregnancy test at Screening
* A male participant must be sexually abstinent (defined as refraining from sexual intercourse from Day 1 (day of dosing) until 90 days after study drug intake) or who is sexually active (either heterosexual, including with a pregnant woman, or homosexual) must agree to use a barrier method of contraception (example, condom) from Day 1 (day of dosing) until 90 days after study drug intake
* Participant must have a body mass index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kilogram per meter^2 (kg/m2), extremes included
* Participant must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic

Exclusion Criteria:

* Participant with a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic insufficiency, renal dysfunction (calculated creatinine clearance below 60 milliliter per minute (mL/min) at Screening using the Cockroft-Gault equation), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers that it could interfere with the interpretation of the study results should exclude the participant
* Participants with abnormal values for either alanine aminotransferase (ALT) or aspartate aminotransferase (AST) (greater than or equal to [>=]1.25 x upper limit of laboratory normal range [ULN])
* Participants with lack of good/reasonable venous access
* Participants with a past history of heart arrhythmias (extrasystoli, tachycardia at rest) or, history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Participants with a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) criteria within 5 years before Screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, methadone, benzodiazepines, and hallucinogens) at Screening and on Day -1 of each treatment period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-53718678 | Up to 72 hour of Post-dose
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma ConcentrationTime Curve From Time 0 to Time of the Last Quantifiable Concentration (AUC [0last]) of JNJ-53718678 | Up to 72 hour of Post-dose
  The AUC (0-last) is the area under the plasma concentration time curve from time 0 to the time of the last measurable non-below quantification limit concentration, calculated by liner-linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-53718678 | Up to 72 hour of Post-dose
  The AUC (0-infinity) is the area under the plasma concentration time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Relative Bioavailability of JNJ-53718678 | Up to 72 hour of Post-dose
  The relative bioavailability based on Cmax, AUC(0last), and AUC(0-inf) will be estimated as 100*Test/Reference, where Test is defined as the pharmacokinetic parameters of oral JNJ-53718678 and Reference is defined as currently existing oral solution G024.
Effect of Food on the Bioavailabilty of JNJ-53718678 | Up to 72 hour of Post-dose
  The effect of food will be evaluated by comparing the pharmacokinetics of JNJ-53718678 under fed conditions with the currently existing oral solution under fasted conditions.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability | Up to 35 days after last study drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium